CLINICAL TRIAL: NCT00930215
Title: Open Label, Randomized, Single Center, 2-way Crossover Bioequivalence Study Comparing Gelatine Capsule 40 mg D961H and HPMC Capsule 40 mg D961H After Repeated Oral Administration in Japanese Healthy Male Subjects
Brief Title: Study Comparing Gelatine Capsule 40 mg D961H and HPMC Capsule in Japanese Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: D961HC00008
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Healthy volunteer; Japanese males; homo-EM; Bioequivalence study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- D961H 40 mg gelatin capsule (Experimental): 2 way crossover
  Interventions: Drug: D961H
- D961H 40 mg HPMC capsule (Experimental): 2 way crossover
  Interventions: Drug: D961H

INTERVENTIONS:
Drug: D961H — Oral gelatin capsule
  Arms: D961H 40 mg gelatin capsule
Drug: D961H — Oral HPMC capsule
  Arms: D961H 40 mg HPMC capsule

SUMMARY:
The purpose of the study is to determine whether the HPMC capsule of D961H 40 mg is bioequivalent to gelatine capsules of D961H 40 mg after a steady state is reached on Day 5

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese
* Classified as homo-EM
* Negative for HIV, Hepatitis B, Hepatitis C and syphilis

Exclusion Criteria:

* Significant clinical illness from 2 weeks preceding the pre-entry visit to the randomization
* Past or present cardiac, renal, hepatic, neurological or gastrointestinal disease

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-06; Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Confirm the HPMC capsule of D961H 40 mg is bioequivalent to the gelatin capsule of D961H 40 mg by assessment of area under the plasma concentration-time curve at steady state on Day 5 | PK sample at Day 5 of treatment period 1 and treatment period 2

SECONDARY OUTCOMES:
Evaluate the PK properties of HPMC capsule of D961H 40 mg following repeated oral doses, by assessment of plasma concentrations, mean residence time, time to maximum plasma concentration and half-life on Day 5 | PK sample on Day 5 of treatment period 1 and treatment period 2
Evaluate the safety and tolerability of HPMC capsule of D961H 40 mg by assessment of AEs, clinical lab tests, ECG, vital signs. | Pre-entry, Day 5 of treatment period 1 and treatment period 2 and follow up (5-7 days after last dose)

CONTACTS AND LOCATIONS:
Overall Officials: Takenobu Masaoka, Study Chair — AstraZeneca; Masataka Date, Study Director — AstraZeneca KK; Shunji Matsuki, Principal Investigator — Kyushu Clinical Pharmacology Research Clinic
Locations (1):
- Research Site, Fukuoka, Japan